CLINICAL TRIAL: NCT03264469
Title: DIAGNOSIS and FORENSIC MANAGEMENT OF PSYCHOLOGICAL TRAUMA IN PATIENTS INVOLVED IN THE TERRORIST ATTACK IN NICE ON THE 14TH JULY 2016
Brief Title: Improvement of the Diagnosis and Medico-legal Management of Psychological Trauma in Patients Involved in the Terrorist Attack in Nice on the 14th July 2016
Acronym: PSYCHIC
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: LOISEAU 2016
Record Dates: First submitted 2017-08-25; First posted 2017-08-29 (Actual); Last update posted 2017-09-19 (Actual); Status verified 2017-09

CONDITIONS: Registration of a Complaint Following the Terrorist Attack of 14 July 2016

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Psychological trauma is a major public health concern that affects numerous patients who have experienced traumatic events.

The objective of our research was to improve the diagnosis and management of persons experiencing such events.

We will seek to determine factors brought into play in the construction of psychological trauma and the best way to identify them so as to implement the optimal management of patients and ensure recognition of this condition.

In addition, in the context of our activity as expert witnesses, we will study the methods used to assess and quantify psychological trauma.

In this respect, a medical appointment will be made by a nurse of the Forensic Medicine Department of Dijon CHU. During this consultation, a self-report questionnaire will be completed by the patient alone to evaluate the level of acute stress followed by a psychiatric consultation and completion of the IES-R questionnaire with the doctor to identify symptoms of psychological trauma.

ELIGIBILITY:
Inclusion Criteria:

- Patients who have registered a complaint leading to the involvement of the Forensic Medicine Department of DIJON CHU to evaluate requests for temporary sick leave for psychological reasons following the event in NICE on the 14 July 2016.

Exclusion Criteria:

* Refusal of the patient to attend the consultation proposed by the Forensic Medicine Department of DIJON CHU,
* Refusal of the patient to take part in a clinical study.
* Verbal information about the clinical study when the appointment was made by the Forensic Medicine nurse,
* Reiteration of the verbal information during the consultation,
* A letter and an official information document given to each patient by the DIJON CHU research Unit stating the objectives and methods of the clinical study,
* Contact details of the Forensic Medicine Department given to patients if they have any questions about the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Registration of a complaint following the terrorist attack of 14 July 2016
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
PID scale | At baseline

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France